CLINICAL TRIAL: NCT04980183
Title: A Clinical Trial of Precise Positioning and Intelligent Operation of Surgical Robots to Reconstruct Cruciate Ligaments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2021156
Record Dates: First submitted 2021-06-25; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Cruciate Ligament Rupture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic surgical robot assisted navigation and positioning for cruciate ligament reconstruction (Experimental): Patient undergoes cruciate ligament reconstruction with robot-assisted navigation and positioning under arthroscopic surgery
  Interventions: Device: Arthroscopic surgical robot
- Conventional arthroscopic cruciate ligament reconstruction (Active Comparator): The patient undergoes conventional arthroscopic cruciate ligament reconstruction
  Interventions: Device: Conventional arthroscopic cruciate ligament reconstruction

INTERVENTIONS:
Device: Arthroscopic surgical robot — The surgeon performs cruciate ligament bone canal positioning and ligament reconstruction with the assistance of an arthroscopic surgical robot
  Arms: Arthroscopic surgical robot assisted navigation and positioning for cruciate ligament reconstruction
Device: Conventional arthroscopic cruciate ligament reconstruction — The surgeon performs conventional arthroscopic cruciate ligament reconstruction surgery without other auxiliary equipment
  Arms: Conventional arthroscopic cruciate ligament reconstruction

SUMMARY:
30 patients with the first rupture of the cruciate ligament were divided into two groups as 1:1. Experimental group will be treated with arthroscopic robot-assisted navigation and positioning for cruciate ligament reconstruction. Control group will be treated with conventional reconstruction. This project is used to verify the advantages of surgical robots assisting surgeons in cruciate ligament reconstruction surgery.

DETAILED DESCRIPTION:
In this study, 30 patients with the first rupture of the cruciate ligament were recruited as the research objects, and the ratio of the experimental group and the control group was 1:1. Patients in the experimental group will be treated with arthroscopic robot-assisted navigation and positioning for cruciate ligament reconstruction, and patients in the control group will be treated with conventional reconstruction. All subjects will undergo CT evaluation and clinical function evaluation. This project is used to verify the advantages of surgical robots assisting surgeons in cruciate ligament reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years old, with closed epiphyses;
2. For the first time, the knee joint is simply ruptured with a cruciate ligament and requires surgical reconstruction; it can be combined with meniscus injury, and the Outerbridge injury score is ≤ II;
3. There is no history of trauma or fracture of the ipsilateral knee joint;
4. The medial collateral ligament or the lateral collateral ligament is not damaged or only slightly damaged (no more than degree I).

Exclusion Criteria:

1. BMI is less than 18.5 or greater than 35 kg/m2;
2. Patients with moderate or severe knee degeneration;
3. Those with limited flexion angle (<120 degrees);
4. Cartilage defect area is greater than 2 cm2 or Outerbridge damage score> Grade II.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
3D-CT compares the position of the tibial canal made by the robot-assisted positioning and the traditional positioning method | Knee CT examinations were performed on patients one week after surgery
  Evaluate the position of the reconstructed tibia canal through 3D-CT using Taukada's method, t / T × 100% was used to evaluate the anteroposterior radial orientation of the tibial tract. Use l / L × 100% to evaluate the orientation of the inner and outer diameters of the tibial tract.
3D-CT compares the position of the femoral canal made by the robot-assisted positioning and the traditional positioning method | Knee CT examinations were performed on patients one week after surgery
  Evaluate the position of the reconstructed femoral canal through 3D-CT according to Bernard and Hertel (BH) quadrant method, l / L × 100% and h / H × 100% are used to evaluate the femoral bone canal positioning.

CONTACTS AND LOCATIONS:
Overall Officials: Yingfang Ao, Prof., Principal Investigator — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing Key Laboratory of Sports Injuries， Beijing, China, Beijing, Beijing Municipality, China